CLINICAL TRIAL: NCT00501761
Title: Social Cognitive Theory and Physical Activity After Endometrial Cancer
Brief Title: Physical Activity After Endometrial Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2004-0454; 1R01CA109919-01 (NIH)
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Healthy Controls; Social Cognitive Theory; Behavioral Intervention; Physical Activity; Exercise Program; Questionnaire
MeSH Terms: conditions — Endometrial Neoplasms; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples 5 times per day for 2 consecutive days.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Endometrial Cancer Survivors
  Interventions: Behavioral: Personalized Exercise Program; Behavioral: Questionnaire
- 2: Healthy Participants: Healthy participants that have no history of invasive cancer.
  Interventions: Behavioral: Questionnaire; Behavioral: Suggested Exercise Program

INTERVENTIONS:
Behavioral: Personalized Exercise Program — Walking up to thirty minutes on most days of the week.
  Groups: 1: Endometrial Cancer Survivors
Behavioral: Questionnaire — Questionnaires regarding physical activity, exercise, and quality of life.
  Other Names: Survey
Behavioral: Suggested Exercise Program — Exercise program performed over 7 days.
  Groups: 2: Healthy Participants

SUMMARY:
Researchers propose to apply Social Cognitive Theory to improve understanding of the mechanisms of physical activity adherence for endometrial cancer survivors participating in a physical activity intervention.

The specific aims of the study are:

1. To test a Social Cognitive Theory-based model of physical activity adoption among sedentary endometrial cancer survivors receiving an intervention to increase physical activity. The model includes hypotheses about the effect of self-efficacy and outcome expectations on physical activity adherence, the effects of four sources of efficacy information (mastery experience, verbal persuasion, modeling, and physiological feedback) on self-efficacy and subsequent exercise adherence, and the influence of physical activity outcomes on subsequent self-efficacy, outcome expectations, and physical activity.
2. To elucidate the influence on self-efficacy of cardiorespiratory fitness and somatic sensations while engaging in physical activity.
3. To determine whether the received dose of an intervention based on Social Cognitive Theory is related to physical activity adherence.
4. To test the effects of adherence to physical activity on endometrial cancer survivors' quality of life and stress as assessed by self-report and salivary cortisol.
5. To test the feasibility of a web-based maintenance intervention for women who have completed the phone counseling portion of the study.

DETAILED DESCRIPTION:
Women who have been successfully treated for endometrial cancer will be invited to participate in the study. After you agree to participate you will be asked questions about your physical activity to make sure you are eligible. You will only be allowed to participate in this study if your physician feels it is safe for you to engage in moderate physical activity, so you will be asked to have him or her complete a form about your health conditions. Information about you cancer and treatment history will be collected from your medical records as part of the study.

If you agree to take part in this study, you will come to M. D. Anderson for study visits twice at the beginning of the study. If needed, the activities for these first 2 visits can be combined into 1 visit, though it will mean that the single visit will take a little longer than each of the 2 visits. After the first visit, you will be asked to return after 2, 4, and 6 months. Each visit will take about 2 hours. Three (3) months and 6 months after the last visit, you will be called to answer questions about your physical activity. It will take about 10 minutes to answer the questions. In case you cannot be reached by phone, the questionnaires will be mailed to you. You will be asked to mail the questionnaire back in with a pre-paid addressed envelope.

At the first visit you will complete questionnaires about your quality of life, medical conditions, and how physically active you are currently and have been in the past. The questionnaires will take about 45 minutes to complete. A baseline electrocardiogram (ECG-a test to measure the electrical activity of the heart) will be performed. If your ECG test is not normal you will be informed. You will practice using the exercise bicycle that will be used in the fitness testing at the later visits. You will be asked to provide a saliva sample by placing a cotton roll in your mouth until it is saturated and then placing it back in a plastic vial without using your hands. This sample will be for practice and will be discarded.

You will also be given an ActiGraph to wear for 5 days. This is a small light device that you wear on your waist during the day. It records how active you are. You will also be given a handheld computer that you will use for 5 days to answer questions about physical activity. The computers are small (about 4-1/2 by 3 inches) and light (about 4 1/2 ounces). The computer will prompt you to enter information up to 8 times a day. Answering these questions will take up to 5 minutes. You will be asked to return the Actigraph and the computer on your second visit.

After 5 days, you will come back to M. D. Anderson for your second study visit. During this visit, you will be asked to complete questionnaires about physical activity that will take about 1 hour. You will have an electrocardiogram (ECG--a test to measure the electrical activity of the heart) performed. You will perform a fitness test, in which you will ride a stationary bicycle while your heart rate, blood pressure, and respiration (breathing) are monitored. You will also be asked to complete two tasks on a computer. After the second visit, you will again use the handheld computer and wear an Actigraph for 5 days. You will also be given 10 vials with a container bag and instructions on collecting saliva samples. You will be asked to provide saliva samples 5 times per day for 2 consecutive days.

During your second visit, you will meet with an exercise physiologist, a specially-trained health care professional who will design a personalized exercise program for you, that will involve walking (up to 30 minutes) on most days of the week. If walking is difficult or painful for you, another form of exercise will be substituted. In addition to receiving a personalized exercise program, you will also receive telephone counseling between your visits to M. D. Anderson and printed materials. Both will provide information and support for your exercise program. The telephone counseling calls will take place once a week during the first 2 months, every other week during Months 3 and 4, and once a month during Months 5 and 6. The phone counselor will talk to you about your exercise program and how it is working for you. The telephone calls will take place at a time that is convenient to you, and will take about 15-20 minutes each time. Some of these telephone counseling calls may be audiotaped, so that the counselors' supervisors can make sure the counseling is done correctly.

During each of the 2-month, 4-month, and 6-month clinic visits (Visits 3, 4, and 5), you will do another fitness test, and any necessary adjustments to your exercise program will be made. This means that if the goals for exercise were set too high or too low, how often the exercise occurs or how long each exercise session lasts will be changed. For example, if the exercise physiologist first recommended that you walk for 15 minutes a day 5 days a week, but you report that you can't walk for 15 minutes, the length of the walk may be reduced. You will also fill out the questionnaires and do the tasks on the computer at these visits. You will complete a brief (5 minutes) program evaluation. You will also be asked to answer questions on the handheld computer for 5 days before and after each these visits. You will also be asked to wear the Actigraph for 5 days before and after each of these visits. At the last visit, you will also be given 10 vials with a container bag and instructions on collecting saliva samples. You will be asked to provide saliva samples 5 times per day for 2 consecutive days. The study staff will give you a prepaid mailing envelopes so you can return the computer, the Actigraph, and the package of vials to them by mail, after the last 5-day period.

This is an investigational study. Up to 326 participants will be enrolled for this study. For the pilot phase, which has been completed, 22 endometrial cancer survivors and 37 comparison participants with no history of cancer were enrolled. For the main phase of the study, for which you are enrolling, up to 267 endometrial cancer survivors will be enrolled. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Survivor of endometrial cancer (survivor group only).
2. Was diagnosed with Stage I, II, or IIIa endometrial cancer in the past five years (survivor group only).
3. Completed surgical or radiation treatment at least 6 months ago (survivor group only).
4. No history of invasive cancer, except for non-melanoma skin cancer (no cancer history group).
5. Age 45 years of older (no cancer history group).
6. Female (no cancer history group).
7. Not pregnant by self-report (no cancer history group).
8. Speaks and reads English (all participants).
9. Oriented to person, place, and time (all participants).
10. Has clearance from their physician to engage in moderate physical activity (all participants).
11. For web-based maintenance intervention pilot study, women will be included if they have completed their third follow-up assessment.
12. For web-based maintenance intervention, women are considered ineligible if they do not have internet access.

Exclusion Criteria:

1. Engages in programmatic physical activity at moderate or greater intensity on five or more days per week for 30 minutes or more, or vigorous intensity activity 20 minutes or more at least 3 days per week, and have maintained this level of activity for six months or longer.
2. Have any condition defined by the American College of Sports Medicine's as "absolute contraindications to exercise testing" (a recent significant change in the resting ECG suggesting significant ischemia, recent myocardial infarction (within 2 days) or acute cardiac event; unstable angina; uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise; severe symptomatic aortic stenosis; uncontrolled symptomatic heart failure; acute pulmonary embolus or pulmonary infarction; acute myocarditis or pericarditis; suspected or known dissecting aneurysm; acute infection).
3. Have any condition as defined by the American College of Sports Medicine's as "relative contraindications to exercise testing" (left main coronary stenosis; moderate stenotic valvular heart disease; electrolyte abnormalities; severe arterial hypertension at rest; hypertrophic cardiomyopathy and other forms of outflow tract obstruction; neuromuscular, musculoskeletal, or rheumatoid disorders that are exacerbated by exercise; high-degree atrioventricular block; ventricular aneurysm; uncontrolled metabolic disease; chronic infectious disease).
4. Right or left bundle branch block.
5. Baseline ST segment or T wave changes that would make monitoring of the ECG stress test indeterminate.
6. Uncontrolled asthma
7. Have other medical contraindications as defined by the patient's physician.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants that have survived endometrial cancer and healthy participants that have no history of invasive cancer.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Estimated)
Dates: Start 2005-05 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Physical activity adoption and adherence in endometrial cancer survivors | Assessments will take place every 2 months, for 4 assessments over a 6-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Robertson MC, Lyons EJ, Song J, Cox-Martin M, Li Y, Green CE, Pinto BM, Carmack CL, Harrison C, Baum G, Basen-Engquist KM. Change in physical activity and quality of life in endometrial cancer survivors receiving a physical activity intervention. Health Qual Life Outcomes. 2019 May 27;17(1):91. doi: 10.1186/s12955-019-1154-5. PMID 31133040
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org